CLINICAL TRIAL: NCT03745261
Title: A Multi-center, Open-label, Randomized, Controlled Study to Evaluate the Effectiveness of Yong Chong Cao Capsule on Outcomes in Patients With Mild to Severe COPD
Brief Title: Effect of Yong Chong Cao Capsule on Outcomes in Patients With Mild to Severe COPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yong Chong Cao for COPD
Record Dates: First submitted 2018-11-15; First posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; mild, moderate, severe; Medicine, Chinese Traditional; Cordyceps sinensis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lymphoma, Follicular | interventions — Albuterol; Tiotropium Bromide; Salmeterol Xinafoate; Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YCC capsule+conventional medicine (Experimental): Patients in this group will be given Yong Chong Cao (YCC) capsule and conventional medicine based on the classes of medications recommended by 2017 GOLD and Chinese Treatment Guidelines for COPD,which are Group A patients: Salbutamol (Ventolin®),Group B and Group C patients: Tiotropium Bromide (Spiriva®),Group D patients: Salmeterol / fluticasone (Seretide®).
  Interventions: Drug: Salbutamol (Ventolin®); Drug: Tiotropium Bromide (Spiriva®); Drug: Salmeterol / fluticasone (Seretide®); Drug: YCC capsule
- BL capsule + conventional medicine (Experimental): Patients in this group will be given Bailing (BL) capsule and conventional medicine based on the classes of medications recommended by 2017 GOLD and Chinese Treatment Guidelines for COPD, which are Group A patients: Salbutamol (Ventolin®),Group B and Group C patients: Tiotropium Bromide (Spiriva®),Group D patients: Salmeterol / fluticasone (Seretide®).
  Interventions: Drug: Salbutamol (Ventolin®); Drug: Tiotropium Bromide (Spiriva®); Drug: Salmeterol / fluticasone (Seretide®); Drug: BL capsule

INTERVENTIONS:
Drug: Salbutamol (Ventolin®) — According to the revised 2017 GOLD, patients will be divided into Group A, B, C, and D based on individualized assessment. Salbutamol will be used to Group A patients: Salbutamol (Ventolin®, GlaxoSmithKline) 100μg/dose. 100 μg each time (when needed), and the maximum dose is 8-12 inhalations a day.
  Other Names: Group A patients: Salbutamol (Ventolin®).
Drug: Tiotropium Bromide (Spiriva®) — Tiotropium Bromide Powder for Inhalation will be used to Group B and Group C patients: Tiotropium Bromide Powder for Inhalation(Spiriva®, Boehringer Ingelheim), 18μg/ capsule, 10 capsules. 18μg each time, once daily.
  Other Names: Group B and C patients: Tiotropium Bromide (Spiriva®)
Drug: Salmeterol / fluticasone (Seretide®) — Salmeterol / fluticasone will be used to Group D patients: Salmeterol / fluticasone (Seretide®, GlaxoSmithKline), 50/250 μg / dose, 60 inhalations. 50/250 μg each time, twice daily.
  Other Names: Group D patients: Salmeterol / fluticasone (Seretide®)
Drug: YCC capsule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi of the lung and kidney will be given Yong Chong Cao (YCC)capsule (Kecai®, Guangdong daguang pharmaceutical group Co., Ltd), 1 g each time, three times a day.
  Arms: YCC capsule+conventional medicine
Drug: BL capsule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi of the lung and kidney will be given Bailing(BL) capsule (Bailing®, Huadong Medicine Co.,Ltd), 1 g each time, three times a day
  Arms: BL capsule + conventional medicine

SUMMARY:
The aim of this study is to evaluate the effectiveness of Yong Chong Cao capsule on outcomes in patients with mild to severe Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
The aim of this study is to compare the effectiveness of two treatments for mild to severe COPD patients: one, Yong Chong Cao capsule treatment and conventional medicine based on 2017 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines; the other, Bailing capsule treatment and conventional medicine.

COPD, with high prevalence, morbidity, mortality and economic burdens, affects millions worldwide. Although many therapies exist and are being developed to relieve symptoms and reduce mortality in COPD, most have only been studied in placebo-controlled efficacy studies in highly selected populations. There are few clinical trials to compare therapeutic alternatives in real world. Furthermore, some randomized controlled trials on Yong Chong Cao capsule, one therapeutic type of Cordyceps sinensis in traditional Chinese medicine (TCM) interventions, especially based on the syndrome of insufficiency of qi of the lung and kidney patterns, have been the certain evidence for showing definite effect for COPD patients. In addition, studies in real world populations of COPD that received different cordyceps sinensis therapies that do have efficacy evidence was found wide variations in care delivery. In short, there is a need to compare the effectiveness of two capsule in patients with mild to severe COPD.

This is a multi-center, open-label, randomized, controlled study to evaluate the effectiveness of Yong Chong Cao capsule for patients with mild to severe COPD compared with Bailing capsule. Following a 14 day run-in period, approximately 240 subjects will be randomly assigned to Yong Chong Cao capsule treatment group, Bailing capsule treatment group for 24 weeks. After the 24 weeks treatment period, subjects in two treatments arms will follow-up 24 weeks. The primary outcome measure is the frequency of exacerbations. The secondary efficacy measures include FEV1, dyspnea (MMRC), exercise capacity(6MWD), quality of life (CAT, SGRQ). Safety will be assessed through the collection of adverse events. There will be a total of 4 study visits (baseline, the 12 and 24 weeks of the treatment, the 24 weeks of follow-up).

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of mild to severe COPD.
* Medically stable.
* Syndrome differentiation belongs to syndrome of insufficiency of qi of the lung and kidney.
* Age between 18 and 80 years.
* With the informed consent signed.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Current respiratory disorders other than COPD (e.g., bronchiectasis, bronchial asthma, tuberculosis, lung fibrosis, pulmonary thromboembolic, diffuse panbronchiolitis, lung cancer).
* Complicated with heart failure (NYHA Class III or IV), or myocardial infarction within six months ,or unstable hemodynamics.
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation).
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study.
* Participating in other trials or allergic to the used medicine.
* Participating in other clinical trials with other interventions in one month.
* Allergic to the used medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-06-20 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
The frequency of exacerbation of COPD | Changes in the frequency of exacerbation at the week 12 and week 24 of the treatment phase, and at the week 24 of the follow-up phase compared with baseline.
  The exacerbation of COPD often results in reduced quality of life, increased rate of lung function decline, increased hospitalization. It is important to assess the changes of exacerbations over time.

SECONDARY OUTCOMES:
Changes in Modified Medical Research Council scale scores | Changes in the mMRC scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using Modified Medical Research Council ( mMRC) scale to assess a patient's level of dyspnea. The MMRC scale is a simple grading system that scored from 0 (less severe) to 4 (severe).
Changes in Forced expiratory volume in one second | Changes in FEV1 at the week 24 of the treatment phase and the week 24 of the follow-up phase compared with baseline.
  Forced expiratory volume in one second (FEV1) is the amount of air that can be exhaled in one second. A positive change from baseline in FEV1 indicates improvement in lung function.
Changes in COPD Assessment Test scores | Changes in the CAT scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the COPD Assessment Test ( CAT) , to assess the impact of COPD on a person's symptom, and how this changes over time.
Changes in Six Minutes Walking Distance | Changes in the 6WMD scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the results of six Minutes Walking Distance (6MWD)Test to assess the exercise tolerance.
Changes in St Georges respiratory questionnaire scores | Changes in the SGRQ scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the St. George's Respiratory Questionnaire(SGRQ), to assess the impact of COPD on a person's life, and how this changes over time.
Changes in clinical COPD questionnaire scores | Changes in the CCQ scores at the week 12 and week 24 of the treatment phase, and the week 24 of the follow-up phase compared with baseline.
  Using the clinical COPD questionnaire (CCQ), to assess the impact of COPD on a person's life, and how this changes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Suyun Li, Doctor, Principal Investigator — The First Affiliated Hospital of HUCM
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li S, Xie Y, Lin L, Wu L, Yu X, Ma Z, Yin Q. The Effectiveness of Yong Chong Cao Capsule in Patients With Mild to Severe COPD: A Multi-Center, Randomized, Active-Controlled Trial. J Evid Based Med. 2025 Dec;18(4):e70091. doi: 10.1111/jebm.70091. Epub 2025 Nov 26. PMID 41295088